CLINICAL TRIAL: NCT05352880
Title: Hypomagnesemia and Its Association With Calcineurin Inhibitors Use in Egyptian Renal Transplant Recipients
Brief Title: Hypomagnesemia and Its Association With Calcineurin Inhibitors Use in Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: magnesium and renal transplant
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Renal Transplantation; Complication
Keywords: hypomagnesemia; renal transplant; calcineurin inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transplant recipients (Experimental): They will be recruited from the Renal Transplantation Clinic at Alexandria Main University hospital
  Interventions: Diagnostic Test: serum magnesium level, FEMg

INTERVENTIONS:
Diagnostic Test: serum magnesium level, FEMg — Blood (serum) for: Magnesium (Mg).Urea, creatinine. Calcium (ca), phosphorus (ph).Sodium (Na), potassium (k), chloride (CL).Fasting blood glucose, cholesterol, triglycerides. Intact PTH, 25OH vitamin D.uric acid, albumin. CBC.
  Trough level of cyclosporine or tacrolimus. ii. Urine for:24 hour urinary: Mg, Ca, Ph, Cl and protein. Spot urine sample to calculate fractional excretion of Mg (FEmg)
  . Detailed history taking, Thorough Systemic physical examination.

SUMMARY:
To assess the prevalence and risk factors of hypomagnesemia and its association with calcineurin inhibitor use among Egyptian renal transplant recipients.

DETAILED DESCRIPTION:
Magnesium (Mg) is the fourth cation in the body and the second most prevalent intracellular cation. Intracellular magnesium concentrations range from 5 to 20 mmol/L; 1-5% of it is ionized, the remainder is bound to proteins.

Extracellular Mg represents only 1% of total body Mg and is mostly found in serum with concentrations ranging between 0.65 to 1.05 mmol/L and in red blood cells. It is present in three states; ionized Mg (55-70%), protein bound Mg (20-30%), and Mg complexed with anions such as bicarbonate or phosphate (5-15%). Ionized magnesium has the greatest biological activity. Magnesium homeostasis is maintained by the intestine, bones and kidneys. It is absorbed in the gut and stored in bone mineral, and excess magnesium is excreted by the kidneys and faeces. The majority of magnesium is absorbed in the small intestine by a passive paracellular mechanism, which is driven by an electrochemical gradient. A minor regulatory fraction of magnesium is transported via the transcellular transporter called transient receptor potential channel melastatin member (TRPM) 6 and TRPM7-members of the long transient receptor potential channel family.

Only about 24-76% of dietary consumed magnesium is absorbed in the gut and the rest is eliminated in the faeces.

Intestinal absorption is not directly proportional to magnesium intake but is dependent mainly on magnesium status. Hypomagnesemia is frequently observed after kidney transplantation, in part to immunosuppressive regimens including calcineurin inhibitors (CNI). The incidence of hypomagnesemia has been reported to be higher among tacrolimus compared to cyclosporine-(CsA) treated patients.

Many other factors influence Mg levels after kidney transplantation such as post-transplantation volume expansion, metabolic acidosis, insulin resistance, decreased gastro-intestinal absorption due to diarrhea, low Mg intake and medications such as diuretics or proton pump inhibitors.

Hypomagnesemia was reported to develop frequently within the first few weeks following transplantation. Hypomagnesemia may persist for several years after kidney transplantation. As observed in the general population, serum Mg levels were inversely correlated with glomerular filtration rate.Hypomagnesemia was associated with a greater decline in allograft function and an increased risk of development of chronic fibrotic lesions andgraft loss for patients with ciclosporin induced nephropathy.

In subjects treated with cyclosporine, Mg supplementation improved renal function, reduced tubular atrophy and interstitial fibrosis and prevented kidney function decline. Mg supplementation has been shown to exert an effect of preventing renal damage by using several mechanisms, including innate immune pathways. Indeed, Mg supplementation inhibits monocyte and macrophage recruitment by abolishing expression of chemoattractant proteins (osteopontin and monocyte chemo attractant protein-1), fibrogenic molecules and extracellular matrix proteins. Moreover, Mg induces down-regulation of endothelin-1 expression. Hypomagnesemia has been shown to play a role in the pathogenesis of arterial hypertension, endothelial dysfunction, dyslipidemia and inflammation leading to coronary heart disease (CHD). Low intracellular Mg levels lead to significantly impaired endothelial function together with decreased endothelial NO synthase expression.

ELIGIBILITY:
Inclusion Criteria:

* Duration more than one year after transplantation.
* Serum creatinine less than 2.5 mg/dL.

Exclusion Criteria:

1. Serum creatinine more than 2.5 mg/dL.
2. Patients on diuretics.
3. Patients on magnesium supplementation.
4. Patients with diabetes mellitus.
5. Chronic alcoholism.
6. Patients on proton pump inhibitors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
decrease in serum magnesium | one month
  serum magnesium below normal values

SECONDARY OUTCOMES:
risk factors of hypomagnesemia | one month
  odds ratio of developing hypomagnesemia

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; montasser M Zeid, MD, Study Chair — professor; Iman E El Gohary, MD, Study Chair — professor; shady Fouad Abouelnaga, MD, Study Chair — fellow; Fathyia A Elian, MBBCh, Study Chair — resident
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Jahnen-Dechent W, Ketteler M. Magnesium basics. Clin Kidney J. 2012 Feb;5(Suppl 1):i3-i14. doi: 10.1093/ndtplus/sfr163. PMID 26069819
- [Background] Konrad M, Schlingmann KP, Gudermann T. Insights into the molecular nature of magnesium homeostasis. Am J Physiol Renal Physiol. 2004 Apr;286(4):F599-605. doi: 10.1152/ajprenal.00312.2003. PMID 15001450
- [Background] de Baaij JH, Hoenderop JG, Bindels RJ. Regulation of magnesium balance: lessons learned from human genetic disease. Clin Kidney J. 2012 Feb;5(Suppl 1):i15-i24. doi: 10.1093/ndtplus/sfr164. PMID 26069817
- [Background] Van Laecke S, Van Biesen W. Hypomagnesaemia in kidney transplantation. Transplant Rev (Orlando). 2015 Jul;29(3):154-60. doi: 10.1016/j.trre.2015.05.002. Epub 2015 May 7. PMID 26001746
- [Background] Nijenhuis T, Hoenderop JG, Bindels RJ. Downregulation of Ca(2+) and Mg(2+) transport proteins in the kidney explains tacrolimus (FK506)-induced hypercalciuria and hypomagnesemia. J Am Soc Nephrol. 2004 Mar;15(3):549-57. doi: 10.1097/01.asn.0000113318.56023.b6. PMID 14978156
- [Background] Stevens RB, Lane JT, Boerner BP, Miles CD, Rigley TH, Sandoz JP, Nielsen KJ, Skorupa JY, Skorupa AJ, Kaplan B, Wrenshall LE. Single-dose rATG induction at renal transplantation: superior renal function and glucoregulation with less hypomagnesemia. Clin Transplant. 2012 Jan-Feb;26(1):123-32. doi: 10.1111/j.1399-0012.2011.01425.x. Epub 2011 Mar 14. PMID 21401720
- [Background] Rodrigues N, Santana A, Guerra J, Neves M, Nascimento C, Goncalves J, da Costa AG. Serum Magnesium and Related Factors in Long-Term Renal Transplant Recipients: An Observational Study. Transplant Proc. 2017 May;49(4):799-802. doi: 10.1016/j.transproceed.2017.01.070. PMID 28457398
- [Background] Paravicini TM, Yogi A, Mazur A, Touyz RM. Dysregulation of vascular TRPM7 and annexin-1 is associated with endothelial dysfunction in inherited hypomagnesemia. Hypertension. 2009 Feb;53(2):423-9. doi: 10.1161/HYPERTENSIONAHA.108.124651. Epub 2008 Dec 22. PMID 19103997
- [Background] Ahmadi F, Naseri R, Lessan-Pezeshki M. Relation of magnesium level to cyclosporine and metabolic complications in renal transplant recipients. Saudi J Kidney Dis Transpl. 2009 Sep;20(5):766-9. PMID 19736470
- [Background] Pham PC, Pham PM, Pham SV, Miller JM, Pham PT. Hypomagnesemia in patients with type 2 diabetes. Clin J Am Soc Nephrol. 2007 Mar;2(2):366-73. doi: 10.2215/CJN.02960906. Epub 2007 Jan 3. PMID 17699436